CLINICAL TRIAL: NCT02178384
Title: An In-vivo Study to Evaluate Three Methods of Managing the Distribution of Loading Forces in Mandibular Distal-extension Prostheses (Class I Kennedy's Classification)
Brief Title: Management of Loading Forces Distribution in Mandibular Distal-extension Prostheses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UDDS-RemPro-01-2014
Record Dates: First submitted 2014-06-27; First posted 2014-06-30 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2015-10

CONDITIONS: Mandibular Distal-extension Prostheses
Keywords: Loading Forces; Removable partial dentures; Bilateral distal extension
MeSH Terms: interventions — Denture Precision Attachment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Altered-cast technique (Experimental): Removable partial dentures will be made using altered-cast technique for free saddles.
  Interventions: Procedure: Altered cast technique
- Precision attachments (Active Comparator): Removable partial dentures will be made using precision attachments which will be located on the distal abutment teeth.
  Interventions: Device: Precision Attachments
- Resilient layer (Active Comparator): Removable partial dentures will be made using a resilient-layer on the distal extension of each appliance.
  Interventions: Procedure: Resilient layer

INTERVENTIONS:
Procedure: Altered cast technique — This techniques deals with the procedures that are employed when constructing the removable partial denture on working casts.
  Other Names: Modified case technique
  Arms: Altered-cast technique
Device: Precision Attachments — These are minor attachments used to split the loading forces during appliance wear
  Other Names: Joint Attachments
  Arms: Precision attachments
Procedure: Resilient layer — This is a layer beneath the appliance which helps in reducing the transmission of loading forces to the underlying soft tissues
  Other Names: Flexible layer
  Arms: Resilient layer

SUMMARY:
The two structures that support a mandibular distal extension removable partial denture differ markedly in their visco-elastic response to loading. The difference between the resilience of the residual ridge tissues and the teeth permitted by the periodontal ligament presents a disparity of support that is in contrast to the uniform support accorded a tooth-supported removable partial denture. Hence the denture tends to rotate about its most distal abutments, inducing heavy torsional stresses on alveolar ridges.

Many methods have been used to control this movement, some of them:

1. Implant support on distal extension removable.
2. Stress breakers provide a mean of interposing a flexible connection between the tooth-borne retainer portion of removable partial denture and its distally extended tissue-borne segment.
3. Altered-cast technique.
4. Design development by using mesial indirect retainers rather than distal ones.

The purpose of this study is: (1) to compare bone absorption around abutment teeth nearby the free saddle; (2) denture displacement and pressure on the soft tissue under the denture base of distal extension RPD (Removable Partial Denture) (3) cellular changes in the soft tissue under the denture base of distal extension RPD.

DETAILED DESCRIPTION:
Removable partial dentures (RPD) have an essential role in treating partly edentulous. patients with large toothless spaces, or without posterior dental support (Kennedy Class I).

Rehabilitation with Distal-Extension Removable Partial Denture (DERPD) deserves special attention because of the difference in resilience between the remaining mucosa of the edentulous area and the periodontal ligament of the abutment tooth. When occlusal forces affect the bases, the difference in resilience between the mucosa of the edentulous area and the periodontal ligament of the abutment teeth creates a rotating movement whose axis is located on the occlusal rests on the abutment teeth. This may induce horizontal forces and mainly lateral forces upon them, causing inflammation, gingival retraction, increase in dental mobility and distal residual ridge resorption. This movement may cause a reduction in function, discomfort and trauma to the RPD supporting tissues.

MATERIAL AND METHODS:

Patients will be recruited from the Department of Prosthodontics at the University of Damascus Dental School. Thirty patients will be randomly divided into three groups (A, B, and C). A mandibular bilateral distal-extension removable partial denture will be used for patients in all groups. But every group will have its own specific method of distributing loading forces.

In Group A: A Removable partial dentures will be made by using altered-cast technique for free saddle.The investigators will make a primary impression using stock tray. This will be followed by a final impression by individual tray. After metal framework try-in, ridge regions are removed from uncorrected master cast with saw. Then, corrective impression of ridges will be obtained with soft ZOE impression paste. Therefore, a metal framework with associated corrective impression will be repositioned on tooth portion of master cast prior to altering distal-extension bases.

In Group B: Removable partial dentures will be made by using precision attachments which will be located on the last abutment tooth. At first, crowns will be prepared to receive the precision attachment, then these are cemented to their respective abutment teeth. So that a mean of interposing a flexible connection between the tooth-borne retainer portion of a removable partial denture and its distally extended tissue-borne base will be provided.

In Group C: Removable partial dentures will be made by using resilient-layer in the distal extension of the removable partial denture.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral distal extension in the mandible (Class I Kennedy's Classification).
* Stable systemic health, including absence of a history of cardiovascular disease.
* No evidence of infection or trauma in the oral region.
* Negative history of syndromes or temporomandibular disorders and parafunction.

Exclusion Criteria:

* Other Classes of Kennedy's Classification
* Patients with ages beyond the accepted age range.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-06; Primary Completion 2015-07 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Soft-tissue vertical displacement (STVD) | This variable will be measured at one month, three months and six months following appliance first delivery
  Soft tissue vertical displacement will be measured using an impression technique at the free end saddles.

SECONDARY OUTCOMES:
Bone absorption of abutment teeth | This variable will be measured at one month, three months and six months following appliance first delivery
  The amount bone absorption will be measured using apical radiography.
Cellular changes of the supporting tissues | This variable will be measured at one month, three months and six months following appliance first delivery
  A brush will be used to have a smear of the underlying soft tissues. Cellular changes will be evaluated microscopically. The changes observed will be analysed quantitatively.

CONTACTS AND LOCATIONS:
Overall Officials: Fadi Alhaji Jnaid, DDS MSc, Principal Investigator — PhD student, Department of Removable Prosthodontics, University of Damascus Dental School, Damascus; Alaa' Salloum, DDS MSc PhD, Study Director — Senior Lecturer, Removable Prosthodontics Department, University of Damascus Dental School, Damascus
Locations (1):
- Department of Removable Prosthodontics, University of Damascus Dental School, Damascus, Rif-dimashq Governorate, Syria

REFERENCES:
- [Background] Pellizzer EP, Ferraco R, Tonella BP, Oliveira BJ, Souza FL, Falcon-Antenucci RM. Influence of ridge type on mandibular distal extension removable partial denture. Acta Odontol Latinoam. 2010;23(1):68-73. PMID 20645647
- [Background] Aydinlik E, Akay HU. Effect of a resilient layer in a removable partial denture base on stress distribution to the mandible. J Prosthet Dent. 1980 Jul;44(1):17-20. doi: 10.1016/0022-3913(80)90039-6. PMID 6991675
- [Background] Kratochvil FJ, Thompson WD, Caputo AA. Photoelastic analysis of stress patterns on teeth and bone with attachment retainers for removable partial dentures. J Prosthet Dent. 1981 Jul;46(1):21-8. doi: 10.1016/0022-3913(81)90129-3. PMID 7024514
- [Background] Holmes JB. Influence of impression procedures and occlusal loading on partial denture movement. 1965. J Prosthet Dent. 2001 Oct;86(4):335-41. doi: 10.1067/mpr.2001.119826. No abstract available. PMID 11677525
- [Background] Igarashi Y, Ogata A, Kuroiwa A, Wang CH. Stress distribution and abutment tooth mobility of distal-extension removable partial dentures with different retainers: an in vivo study. J Oral Rehabil. 1999 Feb;26(2):111-6. doi: 10.1046/j.1365-2842.1999.00345.x. PMID 10080307
- [Background] Leupold RJ, Flinton RJ, Pfeifer DL. Comparison of vertical movement occurring during loading of distal-extension removable partial denture bases made by three impression techniques. J Prosthet Dent. 1992 Aug;68(2):290-3. doi: 10.1016/0022-3913(92)90332-5. PMID 1501177
- [Background] Vahidi F. Vertical displacement of distal-extension ridges by different impression techniques. J Prosthet Dent. 1978 Oct;40(4):374-7. doi: 10.1016/0022-3913(78)90115-4. PMID 359787
- [Background] Saito M, Miura Y, Notani K, Kawasaki T. Stress distribution of abutments and base displacement with precision attachment- and telescopic crown-retained removable partial dentures. J Oral Rehabil. 2003 May;30(5):482-7. doi: 10.1046/j.1365-2842.2003.01092.x. PMID 12752927
- [Background] Tebrock OC, Rohen RM, Fenster RK, Pelleu GB Jr. The effect of various clasping systems on the mobility of abutment teeth for distal-extension removable partial dentures. J Prosthet Dent. 1979 May;41(5):511-6. doi: 10.1016/0022-3913(79)90082-9. PMID 374712